CLINICAL TRIAL: NCT06949241
Title: A Single Cycle of Intravenous Immunoglobulin as Adjuvant to Rituximab in Patients With Pemphigus: A Retrospective Cohort Study at a Tertiary Referral Center
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-31-25-027185
Record Dates: First submitted 2025-04-03; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pemphigus Disease; Rituximab (RTx); Intravenous Immunoglobulin
Keywords: Pemphigus; Rituximab; IVIg; Adverse effect
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- RTX group: Adult patients receiving rituximab and systemic corticosteroids without adjuvant IVIg
- RTX+IVIg group: Adult patients receiving rituximab and systemic corticosteroids with adjuvant IVIg

SUMMARY:
Pemphigus is a critical autoimmune skin condition mediated by pathogenic autoantibodies mainly against desmoglein (Dsg)1 and Dsg3, and is traditionally managed with systemic corticosteroids and immunosuppressants.The revolutionary introduction of rituximab (RTX) has opened up a new era of pemphigus treatment by enabling treatment strategies to specifically target CD20+ B cells.Studies have highlighted the superior efficacy of RTX combined with systemic corticosteroids, making this therapy first-line treatment for pemphigus patients.Currently, the main challenge for pemphigus management is to maximize efficacy while preventing relapses and reducing risks over the course of the disease.

RTX achieves maximum effect typically at 4-8 weeks post-treatment, and is associated with an elevated risk of infection.On the other hand, intravenous immunoglobulin (IVIg), historically employed for the management of refractory pemphigus, is appreciated for its rapid action and lack of added immunosuppressive risk.It has also been shown to induce long-term clinical remission, and continues to serve as a rescue therapy for difficult cases.

While there have been reports on the successful use of RTX and concomitant IVIg for treating refractory pemphigus, there is a lack of extensive research weighing the pros and cons of adding IVIg to the currently recommended RTX regimen (Rheumatoid arthritis protocol, RAP). To investigate the efficacy and safety of this combined therapy, we conducted an retrospective cohort study to evaluate the impact of incorporating IVIg into the RTX and systemic corticosteroid treatment protocol for pemphigus patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' files between January 1st, 2019, and December 31st, 2024 from department of dermatology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
2. with a diagnosis of pemphigus vulgaris or foliaceus in active stage based on guideline indicators, including typical clinical presentation, positive direct immunofluorescence microscopy findings, and/or detection of serum anti-Dsg3 and/or Dsg1 immunoglobin (Ig)G autoantibodies
3. treated with RTX in association with oral corticosteroids
4. with a follow-up of at least 48 weeks after RTX treatment initiation

Exclusion Criteria:

1. with a diagnosis of other variants of pemphigus (e.g., paraneoplastic pemphigus, herpetiform pemphigus, IgA pemphigus);
2. concomitant use of other immunosuppressants (e.g., azathioprine, mycophenolate mofetil, methotrexate)
3. previous administration with IVIg for other indications within 12 weeks

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had a clinical presentation of active pemphigus combined with immunological or pathological evidence, and received rituximab and systemic corticosteroids.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
numbers of patients under disease control | week 4, 8, 12, 24, 36, 48 after treatment
  according to Pemphigus S2 Guideline, patients' new lesions cease to form and established lesions begin to heal
Number of patients with relapses | week 4, 8, 12, 24, 36, 48 after treatment
  according to Pemphigus S2 Guideline，patient who has achieved disease control appears ≥3 new lesions/month that do not heal spontaneously within 1 week, or patient's established lesions extend
Adverse event | week 4, 8, 12, 24, 36, 48 after treatment

SECONDARY OUTCOMES:
peripheral CD19+ cell counts | week 4, 8, 12, 24, 36, 48 after treatment
Serum rituximab concentration | week 4, 8, 12, 24, 36, 48 after treatment
immunoglobulin levels | week 4, 8, 12, 24, 36, 48 after treatment
serum anti-Dsg1 and Dsg3 autoantibody levels | week 4, 8, 12, 24, 36, 48 after treatment
Serum anti-rituximab antibody concentration | week 4, 8, 12, 24, 36, 48 after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China